CLINICAL TRIAL: NCT03495453
Title: Directional Versus Orbital Atherectomy Plaque Modification and Luminal Area Assessment of the Femoro-popliteal Artery Via Intravascular Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-00005
Record Dates: First submitted 2018-03-26; First posted 2018-04-12 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) (Active Comparator): OAS (using CSI device) followed by Inpact Admiral drug coated balloon (DCB)
  Interventions: Device: Percutaneous Revascularization of the Femoropopliteal Arteries using a OAS device
- Medtronic's Hawkone Directional Atherectomy system (DAS) (Active Comparator): DAS (using the Hawkone device) followed by DCB
  Interventions: Device: Percutaneous Revascularization of the Femoropopliteal Arteries using a DAS

INTERVENTIONS:
Device: Percutaneous Revascularization of the Femoropopliteal Arteries using a DAS — Diamondback 360 Peripheral Orbital Atherectomy System (OAS) is a small catheter with a diamond crown. The doctor inserts it at the groin and advances into the leg.The OAS works by spinning around inside the artery to "sand down" the buildup of material along the artery walls while leaving the healthy vessel behind.
  Arms: Medtronic's Hawkone Directional Atherectomy system (DAS)
Device: Percutaneous Revascularization of the Femoropopliteal Arteries using a OAS device — HawkOne Directional Atherectomy System (DAS) also is the small catheter with cutting device. Doctor slowly and smoothly advances it across the blockage in your artery and shaves the plaque from the vessel wall and collects it in the reservoir.
  Arms: CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS)

SUMMARY:
This single center prospective, randomized study will be conducted to investigate plaque removal and luminal gain using CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy System (OAS) (St.Paul, MN) versus Medtronic's Hawkone Directional Atherectomy system (DAS) (Minneapolis, MN) assessed by angiography and Intravascular Ultrasound (IVUS) in patients diagnosed with symptomatic obstructive femoro-popliteal disease will be analyzed. Both devices have received clearance by the Food and Drug Administration (FDA) for use by the label indication.Subjects will be randomized in a 1:1 fashion to receive treatment with either OAS (using CSI device) followed by Inpact Admiral drug coated balloon (DCB) or DAS (using the Hawkone device) followed by DCB. Subjects in both arms will undergo IVUS before and after atherectomy, as well as at the conclusion of the procedure. Clinical data will be collected at baseline, immediately prior to the procedure, during and immediately after the procedures, and within 30 days, 6 and 12 months office visits after the procedure. Data may also be collected at office or hospital visits that are not scheduled but occur up to 12 months after the procedure, if they pertain to treatment related to the obstructive SFA disease. Data to be collected for this study includes demographics, medical history, procedural parameters and follow-up. The study will be conducted at one study center, 90 subjects will be enrolled in the trial with plan to accrue 60 subjects - 30 patients enrolled in the OAS arm and 30 patients enrolled in the DAS arm. The duration of the study is expected to be approximately 2 years from the date of first enrollment (1 year for enrollment of 60 subjects and a year for follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Subject's age ≥ 18 years;
* Subject (or Legal Guardian if applicable) is willing and able to provide consent before any study-specific test or procedure is performed, signs the consent form, and agrees to attend all required follow-up visits.
* Chronic, symptomatic lower limb ischemia defined as Rutherford categories 1-4
* Target lesion(s) located in a superficial femoral or popliteal arteries
* Degree of stenosis ≥70% via Qualitative Comparative Analysis (QCA)
* Total Lesion Length ≥ 80 mm and ≤ 150 mm
* Reference Vessel ≥ 3.0 mm and <6.5mm
* Patent infrapopliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (<50% stenosis) to the ankle or foot with no planned intervention.
* Subject is an acceptable candidate for percutaneous intervention using the OAS or DAS in accordance with their labeled indications and instructions for use

Exclusion Criteria:

* Subjects who have an:
* Previously stented target lesion/vessel.
* Subjects who have undergone prior surgery of the SFA/PA in the target limb to treat atherosclerotic disease.
* Presence of aneurysm in the target vessel.
* Interventional treatment is intended for in-stent restenosis at the peripheral vascular site.
* Target vessel with moderate or severe angulation (e.g., > 30°) or tortuosity at the treatment segment, that precludes safe advancement of the atherectomy device.
* Pre-planned interventional treatment includes planned laser, brachytherapy or atherectomy procedure other than OAS or DAS.
* Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated.
* Known hypersensitivity/allergy to antiplatelet, anticoagulant, thrombolytic medications
* Platelet count <80,000 mm3 or >600,000 mm3 or history of bleeding diathesis.
* Patient has any known coagulation disorder, including hypercoagulability
* Receiving dialysis or immunosuppressant therapy.
* Patient has evidence of intracranial or gastrointestinal bleeding within last 3 months.
* Patient has history of severe trauma, fracture, major surgery or biopsy of a parenchymal organ within past 14 days,
* Female patient who is pregnant or nursing a child,
* Current participation in another investigational drug or device clinical study that has not completed the primary endpoint at the time of randomization/enrollment or that clinically interferes with the current study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anvar Babaev, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) | Medtronic's Hawkone Directional Atherectomy System (DAS)
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) | Medtronic's Hawkone Directional Atherectomy System (DAS) | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Full Range); unit: years] | 70 [67 to 73] | 72 [65 to 77] | 71 [65 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 20 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 30 | 27 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Minimal Luminal Area
Description: To be measured via Intravasular Ultrasound (IVUS) before and after atherectomy
Time Frame: Day 0, Immediately before procedure, immediately after procedure
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) | Medtronic's Hawkone Directional Atherectomy System (DAS)
Number analyzed (Participants) | 29 | 30
mm^2 | 5.8 [4.7 to 8.4] | 4 [2.9 to 6.3]

2. Primary Outcome: Change in Percentage Diameter Stenosis (%DS)
Description: Angiographic measurements of diameter stenosis following atherectomy
Time Frame: Day 0, Immediately before and after procedure
Measure: Mean (Standard Deviation); unit: %DS
Arm/Group | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) | Medtronic's Hawkone Directional Atherectomy System (DAS)
Number analyzed (Participants) | 29 | 30
%DS | 39.5 (14.2) | 69.8 (12.1)

3. Secondary Outcome: Change in Percentage Plaque Volume
Description: To be measured and analyzed via Intravascular Ultrasound (IVUS)
Time Frame: Day 0, Immediately before procedure, immediately after procedure
Measure: Median (Inter-Quartile Range); unit: V/V%
Arm/Group | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) | Medtronic's Hawkone Directional Atherectomy System (DAS)
Number analyzed (Participants) | 29 | 30
V/V% | 66.5 [61.8 to 73.2] | 75.6 [69.9 to 81.8]

ADVERSE EVENTS:
Time Frame: 1 year
Description: regular investigator assessment
Arm/Group | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) | Medtronic's Hawkone Directional Atherectomy System (DAS)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 12/29 | 9/30
Other Adverse Events (participants affected / at risk) | 3/29 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) (N=29) | Medtronic's Hawkone Directional Atherectomy System (DAS) (N=30)
Angina (Cardiac disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
PVD (Vascular disorders) | 1 | 0
HTN (Cardiac disorders) | 1 | 0
AFIB (Cardiac disorders) | 0 | 1
AORTIC STENOSIS (Cardiac disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
PNEUMONIA, COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA, PLEURITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DIABETIS (Endocrine disorders) | 1 | 0
CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
CHF (Cardiac disorders) | 1 | 0
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
STABLE ANGINA (Cardiac disorders) | 1 | 0
CHEST PAIN (Cardiac disorders) | 1 | 0
CAD, CABG (Cardiac disorders) | 1 | 1
CAD PCI (Cardiac disorders) | 1 | 0
CHEST PAIN PCI (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CSI's DIAMONDBACK 360® Peripheral Orbital Atherectomy (OAS) (N=29) | Medtronic's Hawkone Directional Atherectomy System (DAS) (N=30)
PVD (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT03495453/Prot_SAP_000.pdf